CLINICAL TRIAL: NCT04507334
Title: Secondary Rupture of Aortic Aneurysm After EVAR Management
Brief Title: Secondary Rupture of Aortic Aneurysm Post EVAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: ID-RCB/EUDRACT
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-stent rupture of the abdominal aorta is a rare occurrence and with few publications: only 2 multicenter studies and one meta-analysis in 2017 listed this complication As well as a few cases reports This study, the first carried out in France, aims to describe the survival in patients with secondary rupture of the aneurysm despite initial treatment with EVAR.

ELIGIBILITY:
Inclusion Criteria:

* - Patient who had a ruptured aortic aneurysm between 01/01/1993 and 07/31/2020)
* Patients whose aortic aneurysm has been treated with EVAR

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with ruptured aortic aneurysm + EVAR
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
describe survival in patient with secondary rupture aneurysm despite endovascular treatment | 20 years
  mortality describe in the group

SECONDARY OUTCOMES:
Compare survival in patients with rupture secondary aneurysm despite treatment | 20 years
  with endovascular according to:
  * management of secondary rupture of the aneurysm
  * the hemodynamic state on arrival in the center treating
  * the size of the aneurysm sac
2) Explore the risk factors for mortality in study patients | 20 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schlosser FJ, Gusberg RJ, Dardik A, Lin PH, Verhagen HJ, Moll FL, Muhs BE. Aneurysm rupture after EVAR: can the ultimate failure be predicted? Eur J Vasc Endovasc Surg. 2009 Jan;37(1):15-22. doi: 10.1016/j.ejvs.2008.10.011. Epub 2008 Nov 12. PMID 19008129
- [Background] Powell JT, Sweeting MJ, Ulug P, Blankensteijn JD, Lederle FA, Becquemin JP, Greenhalgh RM; EVAR-1, DREAM, OVER and ACE Trialists. Meta-analysis of individual-patient data from EVAR-1, DREAM, OVER and ACE trials comparing outcomes of endovascular or open repair for abdominal aortic aneurysm over 5 years. Br J Surg. 2017 Feb;104(3):166-178. doi: 10.1002/bjs.10430. PMID 28160528
- [Background] Wyss TR, Brown LC, Powell JT, Greenhalgh RM. Rate and predictability of graft rupture after endovascular and open abdominal aortic aneurysm repair: data from the EVAR Trials. Ann Surg. 2010 Nov;252(5):805-12. doi: 10.1097/SLA.0b013e3181fcb44a. PMID 21037436
- [Background] Torsello GB, Klenk E, Kasprzak B, Umscheid T. Rupture of abdominal aortic aneurysm previously treated by endovascular stentgraft. J Vasc Surg. 1998 Jul;28(1):184-7. doi: 10.1016/s0741-5214(98)70214-9. PMID 9685145
- [Background] Alimi YS, Chakfe N, Rivoal E, Slimane KK, Valerio N, Riepe G, Kretz JG, Juhan C. Rupture of an abdominal aortic aneurysm after endovascular graft placement and aneurysm size reduction. J Vasc Surg. 1998 Jul;28(1):178-83. doi: 10.1016/s0741-5214(98)70213-7. PMID 9685144
- [Background] Fransen GA, Vallabhaneni SR Sr, van Marrewijk CJ, Laheij RJ, Harris PL, Buth J; EUROSTAR. Rupture of infra-renal aortic aneurysm after endovascular repair: a series from EUROSTAR registry. Eur J Vasc Endovasc Surg. 2003 Nov;26(5):487-93. doi: 10.1016/s1078-5884(03)00350-2. PMID 14532875
- [Background] Bernhard VM, Mitchell RS, Matsumura JS, Brewster DC, Decker M, Lamparello P, Raithel D, Collin J. Ruptured abdominal aortic aneurysm after endovascular repair. J Vasc Surg. 2002 Jun;35(6):1155-62. doi: 10.1067/mva.2002.123758. PMID 12042725